CLINICAL TRIAL: NCT03558711
Title: PSMA-PET/CT for Prostate Cancer
Acronym: NGP1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AGO/2017/006; 2017-003461-96 (EudraCT Number)
Record Dates: First submitted 2018-02-01; First posted 2018-06-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; biochemical recurrence; 18F-PET imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: intravenous [18F]-PSMA-11
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- study group (Experimental)
  Interventions: Diagnostic Test: 18F-PSMA

INTERVENTIONS:
Diagnostic Test: 18F-PSMA — 18F-PET imaging

SUMMARY:
Prostate cancer is the most frequently occurring male cancer in Belgium. Patients who have been treated for prostate cancer, i.e. by surgery and/or radiotherapy, in a substantial degree suffer from a tumor recurrence, often diagnosed by an increase in serum tumor marker PSA (prostate specific antigen) within the first few years. In these patients with evidence of a tumor recurrence after primary treatment, it is important to most exactly define the location(s) of tumor, to guide appropriate therapy by surgery, radiotherapy and/or hormonotherapy. In so-called oligo-metastatic disease targeted therapy may still be curative and prevent the disease from spreading to distant locations. Therefore it is of paramount importance to have an accurate tool of medical imaging to localize all possible locations to be treated.

With some patients, the PSA-value is so low, that conventional nuclear medicine bone scanning or radiological CT or MRI cannot determine where the metastases are. Therefore, [18F]-Choline PET-CT was introduced to improve diagnostic imaging performance. However, in 30 to 40 percent of patients choline-PET does not localize tumor either, especially in small tumors and/or very low PSA values.

The PSMA PET is already routinely used in many European centres, and has shown a superior accuracy in these patients as compared to conventional imaging techniques. This has been a very consistent finding in scientifically reported patient studies.

Most of these investigations have been performed with PSMA labeled with Gallium-68. The investigators in Ghent, as others, have labeled PSMA with Fluor-18. This tracer provides many advantages, including a higher production yield enabling more patients to be scanned. Also from a perspective of radioprotection and financial costs, Fluor-18 is a better choice. Moreover, several recent studies, comparing Fluor with Gallium modalities seem to suggest equivalent or better diagnostic results, possibly because of a lower aspecific background activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with prostate cancer, either in the setting of diagnosis of biochemical recurrence after curative treatment (prostatectomy with or without lymphadenectomy or radiotherapy), or at primary diagnosis and staging.

Exclusion Criteria:

* Age < 40 or > 70 years in phase-1; upper age limit is not applicable for the phase-2 trial.

Most patients will be > 65 years old, an estimate may be more than 80%.

* Physically or mentally unfit to perform the sequential procedures
* Refusal of patient to be informed about accidental findings on scans.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with prostate cancer
Enrollment: 6 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Safety of administration - follow up of adverse events | Adverse events are followed up until 24 hours after PSMA administration.
  Follow up of treatment-related adverse events according to CTCAE v4.0 criteria.
Safety of administration - change in blood pressure | hourly checking of blood pressure from timepoint of 18F-PSMA-11 injection up to 5 hours post 18F-PSMA injection
  Changes in blood pressure (systolic and diastolic, expressed in mm Hg)
Safety of administration - change in temperature | hourly checking of temperature from timepoint of 18F-PSMA-11 injection up to 5 hours post 18F-PSMA injection
  Changes in temperature (expressed in °C)
Safety of administration - change in heart rate | hourly checking of heart rate from timepoint of 18F-PSMA-11 injection up to 5 hours post 18F-PSMA injection
  Changes in heart rate (expressed in beats per min)
Safety of administration - erythrocytes | before and 300 minutes after 18F-PSMA administration
  Changes in erythrocytes count in plasma (expressed in 10^6/µL)
Safety of administration - haemoglobin | before and 300 minutes after 18F-PSMA administration
  Changes in haemoglobin concentration in plasma (expressed in g/dL)
Safety of administration - leukocytes | before and 300 minutes after 18F-PSMA administration
  Changes in leukocytes count in plasma (expressed in 10^3/µL)
Safety of administration - thrombocytes | before and 300 minutes after 18F-PSMA administration
  Changes in thrombocytes count in plasma (expressed in 10^3/µL)
Safety of administration - sodium | before and 300 minutes after 18F-PSMA administration
  Changes in sodium concentration in serum(expressed in mmol/L)
Safety of administration - creatinine | before and 300 minutes after 18F-PSMA administration
  Changes in creatinine concentration in serum (expressed in mg/dL)
Safety of administration - AST | before and 300 minutes after 18F-PSMA administration
  Changes in AST concentration in serum (expressed in U/L)
Safety of administration - ALT | before and 300 minutes after 18F-PSMA administration
  Changes in ALT concentration in serum (expressed in U/L)
Safety of administration - Alkaline phosphatase | before and 300 minutes after 18F-PSMA administration
  Changes in alkaline phosphatase concentration in serum (expressed in U/L)
Biodistribution of 18F-PSMA | 0 to 300 minutes after 18F-PSMA administration
  Follow up of 18F-PSMA distribution over time in blood, urine, and organs. 18F-PSMA

SECONDARY OUTCOMES:
Establishment of critical organs | 0 to 300 minutes after 18F-PSMA administration
  Based on the biodistribution of 18F-PSMA (primary outcome 14), it will be investigated which organs receive the highest radiation dose (expressed in mGy/MBq).
Investigation of the stability of 18F-PSMA over time in plasma | 0 to 300 minutes after 18F-PSMA administration
  The stability of 18F-PSMA will be assessed via measurement of the percentage defluorination of the compound. Free 18F will be separated from 18F-PSMA using solid-phase extraction, radioactivity (kBq/cc) of each fraction will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- university hospital, Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No